CLINICAL TRIAL: NCT04997031
Title: Tap Water Intake and Perceptions in US Latinx Adults
Acronym: TWIPLA
Status: Completed | Type: Observational
Sponsor: Arizona State University (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00014055
Record Dates: First submitted 2021-07-27; First posted 2021-08-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Latinx Adults 18 - 65 y

SUMMARY:
The purpose of this exploratory cross-sectional investigation is to evaluate associations between tap water perceptions, water consumption behaviors, and hydration status in Latinx adults (18 - 65 y). The objective is to identify perceptual determinants that explain the associations between tap water avoidance and plain water intake and hydration status in Latinx adults.

Aim 1: Characterize the degree to which individual- and community-level factors uniquely predict the perception that tap water is not safe in Latinx adults.

Aim 2: Evaluate household income, education level, and US nativity as potential moderators of the associations between predictors and perceptions of tap water safety.

Aim 3: Evaluate the influence of tap water safety perceptions on plain water intake and 24-h hydration status, after adjustment for predictors of tap water safety perceptions, in a sub-sample of Latinx adults.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Hispanic or Latinx
* English- and/or Spanish-speaking
* Interested in participating in both study phases
* Live in Phoenix, Arizona

Exclusion Criteria:

* Currently pregnant or breastfeeding
* Currently use diuretics
* Do not have access to a desktop, laptop, tablet, or smartphone
* Do not have internet access

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Residents of Phoenix, Arizona
Sampling Method: Non-Probability Sample
Enrollment: 492 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Perception of tap water safety | 1 day
  This will be measured via the question "What is your level of agreement with the following statement: My tap water is safe to drink." Possible responses include strongly disagree, disagree, agree, or strongly agree.
Plain water intake (mL) | 3-day average
24-h urine osmolality (mmol/kg) | 1 day

SECONDARY OUTCOMES:
24-h urine volume (mL) | 1 day
Total water intake (mL) | 3-day average

CONTACTS AND LOCATIONS:
Locations (1):
- Interdisciplinary Science and Technology Building 8, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No